CLINICAL TRIAL: NCT06243848
Title: Comparison of Ultrasound-Guided Injection With Traditional Median Nerve Decompression Surgery in Patients With Carpal Tunnel Syndrome: Randomized Controlled Study
Brief Title: Comparison of Ultrasound-Guided Injection With Median Nerve Decompression Surgery in Carpal Tunnel Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Nuran Eyvaz, Asistant Profesor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTSHDvsOP
Record Dates: First submitted 2024-01-25; First posted 2024-02-06 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Musculoskeletal Diseases; Median Nerve Disease; Carpal Tunnel Syndrome; Ultrasound-Guided Injection; Surgery
Keywords: Carpal Tunnel Syndrome; Ultrasound-Guided Injection; Median Nerve Decompression
MeSH Terms: conditions — Musculoskeletal Diseases; Median Neuropathy; Carpal Tunnel Syndrome | interventions — Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimal Incision Surgery for median nerve decompression (Active Comparator): Classic minimal incision surgical technique for median nerve decompression in patients diagnosed with mild, moderate, and severe carpal tunnel syndrome.
  Interventions: Procedure: Minimal Incision Surgery for median nerve decompression
- Ultrasound-guided perineural injection with 5 cc 5% Dextrose (Experimental): The median nerve will be identified using ultrasound at the proximal entrance of the carpal tunnel. Using an ulnar approach with the in-plane technique, it was planned to inject 5 cc of 5% dextrose around the median nerve.
  Interventions: Procedure: Ultrasound-guided perineural injection with 5 cc 5% Dextrose

INTERVENTIONS:
Procedure: Minimal Incision Surgery for median nerve decompression — Classic minimal incision surgical technique for median nerve decompression in patients diagnosed with mild, moderate, and severe carpal tunnel syndrome.
  Arms: Minimal Incision Surgery for median nerve decompression
Procedure: Ultrasound-guided perineural injection with 5 cc 5% Dextrose — The median nerve will be identified using ultrasound at the proximal entrance of the carpal tunnel. Using an ulnar approach with the in-plane technique, it was planned to inject 5 cc of 5% dextrose around the median nerve.
  Arms: Ultrasound-guided perineural injection with 5 cc 5% Dextrose

SUMMARY:
The aim of this study is to compare ultrasound-guided perineural injection of the median nerve with classic minimal incision surgical technique for median nerve decompression in patients diagnosed with mild, moderate, and severe carpal tunnel syndrome.

DETAILED DESCRIPTION:
Carpal tunnel syndrome represents the most prevalent type of entrapment neuropathy. Anatomically, the carpal tunnel is formed by the carpal bones and lies beneath the transverse carpal ligament, housing nine tendon sheaths of the forearm flexors along with the median nerve. From a clinical perspective, individuals with carpal tunnel syndrome typically experience sensory symptoms such as paresthesia and hypoesthesia, as well as motor impairments and pain within the region supplied by the median nerve, all resulting from mechanical compression and localized ischemia.

In the classification of CTS, participants are diagnosed with mild, moderate, or severe CTS, and various treatment options are available for each category. Treatment options aimed at alleviating symptoms include physical therapy, splinting, wrist injections, and surgical procedures Ultrasound-guided injections of peripheral nerves are typically more advantageous than blind injections because minimize the risk of damaging crucial vascular structures in the adjacent tissue alongside the nerves and decrease the likelihood of intraneural injections.

CTS can also be treated surgically, although the literature has not provided sufficient evidence to establish the superiority of one surgical technique over another. However, these procedures are known to be effective by reducing the volume of the carpal tunnel, thereby relieving pressure on the median nerve. In CTS surgery, following a mini-incision, the dissection proceeds through fat and fascial tissue until the flexor retinaculum is reached, ensuring decompression of the median nerve. The advantages of the mini-incision technique include the preservation of neurovascular structures, a low risk of complications, and a high level of patient satisfaction, making it a prominent surgical approach.

The aim of this study is to compare ultrasound-guided perineural injection of the median nerve with the classic minimal incision surgical technique for median nerve decompression in participants diagnosed with mild, moderate, and severe carpal tunnel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* The presence of symptoms such as nocturnal, posture-related, or movement-related paresthesias, along with possible pain, in the area supplied by the median nerve in the hand, lasting for more than 3 months.
* Confirmation of mild, moderate or severe CTS through electrophysiological testing.
* Numbness and loss of sensation in the hand's regions innervated by the median nerve, as well as weakness in the thenar muscles innervated by the median nerve.
* Positive results on either the Phalen test and/or Tinel sign.

Exclusion Criteria:

* Individuals who may exhibit symptoms mimicking carpal tunnel syndrome, such as cervical radiculopathy, polyneuropathy, brachial plexopathy, or thoracic outlet syndrome.
* Patients who have received a previous injection into the carpal tunnel within the past 6 months.
* Thenar muscle atrophy.
* A history of prior carpal tunnel surgery.
* Regular usage of systemic nonsteroidal anti-inflammatory drugs and corticosteroids.
* Pregnancy
* Patients diagnosed with rheumatoid arthritis, systemic lupus erythematosus, gout, systemic sclerosis, dermatomyositis, or polymyositis.
* Malignancy.
* Active infections

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2025-11-24 (Estimated); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
Change from baseline visual analog scale (VAS) wrist pain at 4th and 12th week | baseline and 12th week
  Pain intensity was assessed using a visual analogue scale for pain, ranging from 0 to 10 mm, where 0 indicates the absence of pain and 10 signifies intense pain. This scale is widely recognized for its strong reliability and validity in measuring musculoskeletal pain.

SECONDARY OUTCOMES:
Change from baseline Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) at 4th and 12th week | baseline and 12th week
  The Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) is a commonly used questionnaire for CTS, comprising two main components. It assesses severity using two categories: a symptom severity scale with 11 questions and a functional status scale with 8 questions. Each question is rated on a scale of 0 to 5, where 0 indicates no difficulties during the activity, and 5 indicates extremely severe dysfunction.
Change from baseline Cross-sectional area of the Median Nerve (CSA) at 4th and 12th week | baseline and 12th week
  The median nerve's cross-sectional area (CSA) will be assessed at the scaphoid-pisiform level using an ultrasound. Three measurements will be taken, and the analysis will utilize the average of these three measurements.
  CSA values increase as clinical findings worsen.
Change from baseline Electrophysiological Evaluation at 4th and 12th week | baseline and 12th week
  Antidromic sensory nerve conduction velocity and distal motor latency of the median nerve will be assessed for all patients. These measurements will be performed three times, and the resulting average value will be considered. CTS will be identified as mild, modarate or severe by electrophysiologic evaluations.
Change from baseline Hand Grip Strength Assessment at 4th and 12th week | baseline and 12th week
  The participants' hand grip strength will be assessed using the "Jamar Hydrolic Hand Dynamometer." . Patients will be instructed to exert maximum force, and each measurement will be repeated three times, with the averages recorded in kilograms. Higher scores indicate better grip strength.
Change from baseline Finger Grip Strength Assessment at 4th and 12th week | baseline and 12th week
  Finger grip strength will be evaluated using the "Jamar Digital Pinchmeter." Measurements will be taken bilaterally in three different hand positions: lateral, palmar, and fingertip grips. Higher average scores indicate better finger grip strength. The maximum force exerted during each trial in kilograms will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Nuran EYVAZ, MD, Principal Investigator — Afyonkarahisar Health Sciences University; Ali İzzet AKÇİN, MD, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Afyonkarahisar Health Sciences University, Afyonkarahisar, Turkey (Türkiye)

REFERENCES:
- [Background] Lam KHS, Wu YT, Reeves KD, Galluccio F, Allam AE, Peng PWH. Ultrasound-Guided Interventions for Carpal Tunnel Syndrome: A Systematic Review and Meta-Analyses. Diagnostics (Basel). 2023 Mar 16;13(6):1138. doi: 10.3390/diagnostics13061138. PMID 36980446
- [Background] Lin MT, Liu IC, Syu WT, Kuo PL, Wu CH. Effect of Perineural Injection with Different Dextrose Volumes on Median Nerve Size, Elasticity and Mobility in Hands with Carpal Tunnel Syndrome. Diagnostics (Basel). 2021 May 9;11(5):849. doi: 10.3390/diagnostics11050849. PMID 34065073
- [Background] Pace V, Marzano F, Placella G. Update on surgical procedures for carpal tunnel syndrome: What is the current evidence and practice? What are the future research directions? World J Orthop. 2023 Jan 18;14(1):6-12. doi: 10.5312/wjo.v14.i1.6. eCollection 2023 Jan 18. PMID 36686281